CLINICAL TRIAL: NCT01680484
Title: Bitter Chocolate Versus Orange Juice for Non-reactive Non-stress Test (NST) Patterns: A Randomized Prospective Controlled Study
Brief Title: Bitter Chocolate or Orange Juice for Non-reactive Non-stress Test (NST) Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Sertac ESIN, Principal Investigator, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HEK 10/117-13
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Nonreassuring Fetal Status
Keywords: non-stress test
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Bitter chocolate (Active Comparator): 50 grams Ülker Golden %70 bitter chocolate, İstanbul, Turkey
  Interventions: Dietary Supplement: Bitter chocolate
- Orange juice (Active Comparator): Ülker İçim Orange Juice 250 cc, İstanbul, Turkey
  Interventions: Dietary Supplement: Orange juice
- Control (No Intervention): Sit and rest

INTERVENTIONS:
Dietary Supplement: Bitter chocolate
  Arms: Bitter chocolate
Dietary Supplement: Orange juice
  Arms: Orange juice

SUMMARY:
There are multiple factors affecting the variability and acceleration pattern of fetal heart rate (FHR) pattern. However, fetal activity is considered as the main determinant. Any factor decreasing fetal activity causes a decrease in FHR variability. Fetal activity may be stimulated by manual manipulation, sound, light, change in maternal position and maternal ingestion of glucose. Among those, ingestion of any kind of food or juice is most frequently practiced in outpatient settings. This is not only medical but also a social routine. In this study the investigators have chosen the two most popular so-called 'fetal accelerators', chocolate and orange juice against no intervention and tried to find any usefulness of these on non-reactive NST patterns.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies at 36 to 41 completed gestational weeks that have a non-reactive NST pattern without decelerations.

Exclusion Criteria:

* multiple pregnancies, fetal anomaly, hypertension, intrauterine growth restriction, active labor, contractions or decelerations on NST, absence of a first or second trimester ultrasonography for accurate gestational dating, pre-gestational or gestational diabetes and known allergy to chocolate or orange

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Increase in reactivity of NST | 30 minutes

SECONDARY OUTCOMES:
Increase in the maternal fetal movement perception | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sertac Esin, MD, Principal Investigator — Dr. Sami Ulus Maternity and Children's Training and Research Hospital
Locations (1):
- Dr. Sami Ulus Maternity and Children's Training and Research Hospital, Ankara, Turkey (Türkiye)